CLINICAL TRIAL: NCT05038995
Title: The Effect of Early Cow's Milk Elimination Diet on the Growth Pattern and Nutritional Status of Preschool Children
Brief Title: The Effect of Early Cow's Milk Elimination Diet on the Growth Pattern
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nazlı ERCAN, Principle investigator, Saglik Bilimleri Universitesi
Other Study IDs: NzlKbr2021
Record Dates: First submitted 2021-08-19; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Cow Milk Allergy
Keywords: Cow milk allergy; Elimination diet; Anthropometry; Growth status
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cow milk elimination group: The CME children will be eligible for the study if they (1) had a diagnosis of CMA by OFC, except children with known anaphylaxis (2) those on a CME diet or a specialized infant formula for at least three months (3) had reintroduced cow's milk for at least three months ago. Children who excluded other foods in addition to cows' milk in the first four years of life for ≥ three months and who currently introduced these foods for at least ≥ three months will be also enrolled in the CME group.
- Healthy group: Healthy children will ve eligible for the study if they (1) did not have CMA and other allergic diseases (2) who had never been on a diet throughout their lives.

SUMMARY:
This study aimed to survey the growth of children who were on elimination diet due to cow milk allergy in Turkey. 0-5 year aged children diagnosed with cow's milk allergy (CMA) and healthy age-sex-matched children as the control group was planned for inclusion. Participants will be included in the study by consecutive sampling. The anthropometry measurements (height-for-age [HFA], weight-for-age [WFA], and weight-for-height [WtHt]) will be evaluated according to the Z-score using the WHO ANTHRO [Z-score = Patient's value - Average value / Standard Deviation (SD)]. The Z-score (SDS) in the average child by age was "0".

DETAILED DESCRIPTION:
0-5 year aged children diagnosed with cow's milk allergy (CMA) and healthy age-sex-matched children as the control group was planned for inclusion. The study will constitute of two groups; group 1; the children who received cow's milk elimination (CME) diet and group 2; the healthy controls. Group 1 will constitute of children aged 0-5 years who received a CME diet due to CMA (Ig E-mediated and/or non-Ig E-mediated and/or mixed type)], confirmed by an oral food challenge test (OFC) and had reintroduced cow's milk for at least ≥ three months ago. Participants will be included in the study by consecutive sampling. The anthropometric measurements (height-for-age [HFA], weight-for-age [WFA], and weight-for-height [WtHt]) will be evaluated according to the Z-score using the WHO ANTHRO [Z-score = Patient's value - Average value / Standard Deviation (SD)]. The Z-score (SDS) in the average child by age was "0".

ELIGIBILITY:
Study Group Inclusion Criteria:

* had a diagnosis of CMA by OFC, except children with known anaphylaxis
* those on a CME diet or a specialized infant formula for at least three months
* had reintroduced cow's milk for at least three months ago.
* Children who excluded other foods in addition to cows' milk in the first four years of life for ≥ three months and who currently introduced these foods for at least ≥ three months were also enrolled in the CME group.

Healthy group inclusion criteria:

* did not have CMA and other allergic diseases
* who had never been on a diet throughout their lives.

Exclusion Criteria:

* Known acute (e.g., influenza) or chronic (e.g., diabetes, immune deficiencies ) diseases,
* history of systemic steroid use > 0.5 mg/kg for more than one week in their life,
* recurrent infections within the last three months,
* food restriction other than food allergy (e.g., vegan, vegetarian),
* moderate to severe asthma, and other medical or surgical conditions which might affect nutrition and growth.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric Allergy Department Outpatient Clinic and Healthy Child Outpatient Clinic
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Body weight in kilograms-T0 | One month prior to the diagnosis of CMA
  Body weight (kg)
Body weight in kilograms-T1 | On the 3-month of CME diet
  Body weight (kg)
Body weight in kilograms-T2 | Three months after the end of the CME diet
  Body weight (kg)
Body weight in kilograms-T3 | The last examination date of the patient after 3rd month control after CME diet
  Body weight (kg)
Height in centimeters-T0 | One month prior to the diagnosis of CMA
  Height (cm)
Height in centimeters-T1 | On the 3-month of CME diet
  Height (cm)
Height in centimeters-T2 | Three months after the end of the CME diet
  Height (cm)
Height in centimeters-T3 | The last examination date of the patient after 3rd month control after CME diet
  Height (cm)
Head circumference in centimeters-T0 | One month prior to the diagnosis of CMA
  Head circumference (cm)
Head circumference in centimeters-T1 | On the 3-month of CME diet
  Head circumference (cm)
Head circumference in centimeters-T2 | Three months after the end of the CME diet
  Head circumference (cm)
Head circumference in centimeters-T3 | The last examination date of the patient after 3rd month control after CME diet
  Head circumference (cm)

SECONDARY OUTCOMES:
Dietary intake | The last examination date of the patient after 3rd month control after CME diet
  Three day dietary record
Blood measurements-Hemoglobin | The last examination date of the patient after 3rd month control after CME diet
  Hemoglobin g/dl
Blood measurements-Sodium | The last examination date of the patient after 3rd month control after CME diet
  sodium mg/ml
Blood measurements-Potassium | The last examination date of the patient after 3rd month control after CME diet
  Potassium
Blood measurements-Albumin | The last examination date of the patient after 3rd month control after CME diet
  Albumin
Blood measurements-Protein | The last examination date of the patient after 3rd month control after CME diet
  Protein
Blood measurements-Calcium | The last examination date of the patient after 3rd month control after CME diet
  Calcium
Blood measurements-Vitamin B12 | The last examination date of the patient after 3rd month control after CME diet
  Vitamin B12
Blood measurements-selenium | The last examination date of the patient after 3rd month control after CME diet
  Selenium
Blood measurements-zinc | The last examination date of the patient after 3rd month control after CME diet
  Zinc
Blood measurements-25-OH vitamin D | The last examination date of the patient after 3rd month control after CME diet
  25-OH vitamin D
Blood measurements-iron | The last examination date of the patient after 3rd month control after CME diet
  Iron
Blood measurements-Folate | The last examination date of the patient after 3rd month control after CME diet
  Folate

CONTACTS AND LOCATIONS:
Overall Officials: Nazli Ercan, MD, Principal Investigator — University of Health Sciences Turkey, Gulhane Education and Research Hospital
Locations (1):
- University of Health Sciences, Gulhane Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30412327/